CLINICAL TRIAL: NCT00097474
Title: The Effects of Hydrocortisone, Melatonin, and Placebo on Symptoms of Jet Lag
Brief Title: Effects of Hydrocortisone, Melatonin, and Placebo on Jet Lag
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050037; 05-CH-0037
Record Dates: First submitted 2004-11-23; First posted 2004-11-24 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-05-28

CONDITIONS: Jet Lag
Keywords: Cortisol; Jet Lag; Healthy Volunteer; HV
MeSH Terms: conditions — Jet Lag Syndrome | interventions — Hydrocortisone; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Combination (Experimental): Both HC 30 and ML 5 will be administered
  Interventions: Drug: Hydrocortisone; Drug: Melatonin
- Hydrocortisone (Experimental): 30mg Hydrocortisone will be administered
  Interventions: Drug: Hydrocortisone
- Melatonin (Experimental): 5 mg Melatonin will be administered
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone will be given alone or in combination with Melatonin to see if symptoms of jet lag are alleviated
  Arms: Combination; Hydrocortisone
Drug: Melatonin — Melatonin will be given alone or in combination with Hydrocortisone to see if symptoms of jet lag are alleviated
  Arms: Combination; Melatonin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will examine the effects of cortisol (hydrocortisone), melatonin, a combination of cortisol and melatonin, and placebo (an inactive substance) on jet lag symptoms. Jet lag is a term used to describe symptoms people commonly experience after rapid travel across several time zones. The cause of jet lag is not known, but various hormones, including cortisol and melatonin, have a day-to-night pattern of secretion and play a role in maintaining the body's internal rhythms. This study will test whether taking cortisol, melatonin, or both can help re-establish the body's day-night cycle and result in less jet lag.

People between 18 and 65 years of age who are planning a non-stop eastward flight with the following characteristics may be eligible for this study:

* Crossing six to eight time zones (6 to 8 hours difference between Eastern Standard Time and the destination)
* Destination between 30 and 50 latitudes (approximately Cairo to London)
* Evening flight (5 PM to midnight) with morning arrival
* Remaining abroad at least 4-10 days

Candidates must have a body mass index (BMI) between 20 and 30 kg/M (not too thin and not overweight) and must not be taking medicines that affect sleep or cortisol or melatonin levels. Prospective participants are screened with a medical history, blood tests, and check of blood pressure, height, and weight.

Pre-flight Procedures

Participants keep a sleep journal 3 days before the flight. For 1 day within 3 days of the flight they fill out jet lag and sleepiness questionnaires and collect morning and bedtime saliva samples for measurement of cortisol and melatonin. The saliva is collected by chewing on two small cotton pads and spitting them into a tube. Premenopausal women provide a urine sample the week before the flight to test for pregnancy. On the day of the flight, the participants do not collect saliva or fill out sleep logs or questionnaires. They are given two bottles with study medication. One bottle, labeled "AM," contains either hydrocortisone or placebo; the other, labeled "PM," contains either melatonin or placebo.

Post-flight Procedures

Upon arriving at their destination in the morning, participants obtain a saliva sample and take one of the capsules in the "AM" bottle. At bedtime, they collect saliva and then take one of the "PM" capsules. They repeat the medication doses for a total of 4 days and repeat the saliva collections on days 2 through 4, 7 and 10 after arrival. In addition, participants complete jet lag and sleep questionnaires in the morning, afternoon, and just before bedtime on the day of arrival and on days 2 through 4, 7 and 10.

After they return from their trip, participants are seen at the NIH Clinic to bring in their saliva specimens and review their questionnaires with study investigators.

DETAILED DESCRIPTION:
Jet lag resulting from rapid flight across several time zones is a common complaint of travelers. The symptoms of jet lag are primarily described as daytime sleepiness, fatigue, and impaired mental efficiency and can also include weakness and irritability. It is considered to be due to the desynchronization between the internal circadian rhythm and the new local day-night cycle at the traveler s destination. A means of rapidly resynchronizing the circadian rhythm to the local time would benefit people who suffer severely from this syndrome.

What actually underlies jet lag is a question that has not been fully answered. Various endogenous hormones, including cortisol and melatonin, have a natural circadian rhythmicity and play a role in maintaining the body s internal clock. Cortisol is produced by the hypothalamic- pituitary-adrenal axis in a circadian manner and in response to stress. Normal cortisol has a diurnal rhythm with a maximum level in the morning and a nadir during the night. While a time shift does not change the total daily amount of cortisol that is secreted, the temporal organization of the cortisol secretions is disrupted and the circadian rhythm does not re-entrain for several days. Thus, the first few mornings in a new time zone can be considered relatively cortisol-deficient because the traveler does not experience the peak of cortisol at the time of awakening. Taking exogenous glucocorticoids at the proper time may help re-entrain the circadian rhythm faster and result in less jet lag.

Melatonin is a hormone that is secreted nocturnally by the pineal gland. Exposure to bright light diminishes its release while darkness triggers it. A recent meta-analysis has shown that taking melatonin can alleviate symptoms of jet lag.

The aim of the present study is an attempt for the first time to attenuate jet lag symptoms with hydrocortisone, melatonin, a combination of both hydrocortisone and melatonin or placebo.

Forty-eight normal volunteers will be randomized in blocks of eight to one of four treatment arms: hydrocortisone (25 mg) alone, melatonin (5 mg) alone, hydrocortisone (25 mg) and melatonin (5 mg) in combination, and placebo. Volunteers will travel in an eastwardly direction across 6-8 time zones. Upon morning arrival at the new destination, volunteers will obtain a saliva sample and then take 25 mg hydrocortisone (or placebo). At the target bedtime of (10 pm to midnight local time) they will take 5 mg of melatonin (or placebo). Volunteers will wake up at 7 am-10:30 am (local time) and take 25 mg hydrocortisone (or placebo). Subjects will repeat these dosages for 3 days for a total of four days. Participants also will obtain salivary samples of cortisol and melatonin on awakening and at bedtime on one day before travel and at the new destination for days 1 - 4, 7 and 10 after arrival. The primary outcome measure will be subjective rating of jet lag and components or correlates of this such as fatigue and daytime tiredness. Subjects will keep sleep logs and fill out a symptoms questionnaire daily for 3 days before and 4 days after the flight and on days 7 and 10. Secondary outcomes will be the measurement of salivary cortisol and melatonin. The data obtained from this study will provide an assessment of effective treatment of jet lag syndrome and will provide a better understanding of the role of hormones in the disruption of the circadian rhythm.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18, but less than or equal to 65, male or female.
* Normal physical exam and laboratory results.
* Negative urinary pregnancy test 1 week prior to travel (pre-menopausal women).
* Planned eastward flight crossing 6-8 time zones between 30n and 50n latitudes.
* A minimum stay of 7 - 10 days abroad.
* Willingness and anticipated ability to comply with study procedures, including sleep and wake hours, saliva collection and questionnaire completion.
* Written informed consent.

EXCLUSION CRITERIA:

* BMI less than or equal to 20 or greater than or equal to 30 kg/m.
* Current psychiatric or seizure disorder.
* Current sleep disorder as assessed by presence of sleep apnea, daytime napping of more than 20 minutes, chronic fatigue.
* History of Cushing's syndrome.
* Serious chronic medical condition.
* Current drug or alcohol abuse.
* SGOT or SGPT greater than three-fold normal.
* Current pregnancy or lactation.
* Current use of CPAP.
* Chronic use of beta-blockers (which inhibit melatonin secretion), anti-epileptic agents, anticoagulants, fluvoxamine, nifedipine or soporific or sleep-inducing agents (including benzodiazepines, melatonin), or glucocorticoids.
* Fasting blood glucose greater than 110 mg/dL or known diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-12-21 (Actual); Primary Completion 2006-01-06 (Actual); Study Completion 2007-11-14 (Actual)

PRIMARY OUTCOMES:
improvement in jet lag symptoms | 10 days
  Patients will report jet lag symptoms via questionnaire

SECONDARY OUTCOMES:
salivary cortisol level | 10 days
  salivary cortisol at bedtime will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arendt J, Aldhous M, Marks V. Alleviation of jet lag by melatonin: preliminary results of controlled double blind trial. Br Med J (Clin Res Ed). 1986 May 3;292(6529):1170. doi: 10.1136/bmj.292.6529.1170. No abstract available. PMID 3085768
- [Background] Buxton OM, Copinschi G, Van Onderbergen A, Karrison TG, Van Cauter E. A benzodiazepine hypnotic facilitates adaptation of circadian rhythms and sleep-wake homeostasis to an eight hour delay shift simulating westward jet lag. Sleep. 2000 Nov 1;23(7):915-27. PMID 11083601
- [Background] Cho K, Ennaceur A, Cole JC, Suh CK. Chronic jet lag produces cognitive deficits. J Neurosci. 2000 Mar 15;20(6):RC66. doi: 10.1523/JNEUROSCI.20-06-j0005.2000. PMID 10704520
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-CH-0037.html